CLINICAL TRIAL: NCT00706407
Title: Uro-NIRS Clinical Study
Acronym: Uro-NIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Urodynamix Technologies (Industry); Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0709009413
Record Dates: First submitted 2008-06-02; First posted 2008-06-27 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Lower Urinary Tract Symptoms; Overactive Bladder
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fully integrated Uro-NIRS:UDS (Experimental)
  Interventions: Device: Fully integrated Uro-NIRS:UDS

INTERVENTIONS:
Device: Fully integrated Uro-NIRS:UDS — As part of standard care subjects will be undergoing a standard bladder pressure diagnostic procedure. This standard procedure will involve the insertion of a catheter (a plastic tube) into the urethra and the measurement of pressure within the bladder. For subjects taking part in this study, the health of the bladder will measured by using light instead of pressure. A patch, the size of cell phone or deck of playing cards, will be taped to the skin in the middle of the abdomen, above the bladder. Using laser light that is 300 billion times weaker than the light from a regular household 100-Watt light bulb, the Laborie and Urodynamix device will take measurements through the skin without inserting anything into the body.

SUMMARY:
The purpose of this experiment is to confirm the results of previous testing of Urodynamix's Uro-NIRS device. Together Urodynamix and Laborie have created a device that includes standard Laborie medical equipment and the experimental Urodynamix device. Collectively this integrated device is considered an investigational device, and the results from this study may be used to support a submission to the US Food and Drug Administration for the approval of the integrated device.

This research is being done because we want to test the ability of the integrated Laborie and Urodynamix device to provide a non-invasive method to provide additional information to assist with the diagnosis of or treatment plan of patients suffering from urinary problems. The current technologies rely solely on the measurement of internal pressures of the bladder, which involves the insertion of catheter into the subject's urethra.

DETAILED DESCRIPTION:
This is a study of the fully integrated Uro-NIRS:UDS device (Laborie Triton or Laborie Dorado and Urodynamix's Non-Invasive Urodynamics device - Uro-NIRS), to confirm the results using the fully integrated Uro-NIRS:UDS device as compared to the stand-alone URO-NIRS device and UDS device. The study will evaluate male patients with lower urinary tract symptoms (LUTS) and female subjects with over-active bladder (OAB).

The Uro-NIRS unit uses near infrared light at 3 different wavelengths to measure changes in haemoglobin and cytochrome from the detrusor muscle from the human bladder wall. This process is similar to what is used for cerebral and muscle oxygenation monitoring (e.g., pulse oximetry). Previous clinical feasibility studies have identified the correlation between the changes in haemoglobin and cytochrome and the pressure values obtained during urodynamics procedures and uroflow procedures.

For this study the Uro-NIRS results specifically will not be used by the urologist/nurse to guide in patient management and treatment decisions, but rather will only be used to collect measurements from the patient. The Uro-NIRS sensor patch will be adhered to skin surface where their bladder is located.

The study will be conducted by the two principal investigators at the two clinical study sites who will collectively enrol a minimum of 50 subjects, with a minimum of 35 male subjects and a maximum of 15 female subjects. The study enrolment objective is to equally enrol male subjects into three categories: unequivocal, obstructed and unobstructed. Female subjects shall all have OAB.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older.
* Subjects are patients of one of the institutions and are currently scheduled for UDS
* Male subjects must have LUTS
* Female subjects must have OAB
* Subjects must give their informed consent prior to enrollment.

Exclusion Criteria:

* The patient has an existing health condition which the investigators feel will not allow for safe or accurate measurements with the Uro-NIRS:UDS device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Te, M.D., Principal Investigator — Cornell University
Locations (1):
- New York-Presbyterian Hospital Weill Cornell Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fully Integrated Uro-NIRS:UDS: As part of standard care subjects will be undergoing a standard bladder pressure diagnostic procedure. This standard procedure will involve the insertion of a catheter (a plastic tube) into the urethra and the measurement of pressure within the bladder. For subjects taking part in this study, the health of the bladder will measured by using light instead of pressure. A patch, the size of cell phone or deck of playing cards, will be taped to the skin in the middle of the abdomen, above the bladder. Using laser light that is 300 billion times weaker than the light from a regular household 100-Watt light bulb, the Laborie and Urodynamic device will take measurements through the skin without inserting anything into the body.
Period: Overall Study
Arm/Group | Fully Integrated Uro-NIRS:UDS
Started | 42
Completed | 33
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Obstructed: All patients who had data analyzed
- Unobstructed: Patients with obstruction
- Total: Total of all reporting groups
Arm/Group | Obstructed | Unobstructed | Total
Number analyzed (Participants) | 26 | 7 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Raw data regarding the age of participants in the obstructed group was pooled and not coded. Thus age was not able to be calculated individually, but was reported for the total. | NA (NA) — Raw data regarding the age of participants in the unobstructed group was pooled and not coded. Thus age was not able to be calculated individually, but was reported for the total. | 67 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 7 | 33
Region of Enrollment [Number; unit: participants]
  United States | 26 | 7 | 33
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — International Prostate Symptom Score (IPSS) is a 7 point scale used to screen, track and manage symptoms associated with BPH. The symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Scores range from 1 to 5 for a total of maximum 35 points (0-7 Mildly symptomatic, 8-19 Moderately symptomatic, 20-35 Severely symptomatic)
  units on a scale | 19 (7) | 18 (7) | 19 (7)
Quality of Life (QoL) [Mean (Standard Deviation); unit: units on a scale] — Quality of Life (QoL) is a one point scale used to assess how their symptoms affect their quality of life on the IPSS. A score ranges from 1 to 6, with 6 being the worse outcome.
  units on a scale | 5 (1) | 4 (1) | 4 (1)
Prostate Volume [Mean (Standard Deviation); unit: ml] | 53 (42) | 28 (23) | 48 (39)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/ml] — Prostate Specific Antigen (PSA) is a protein that is produced by the cells in the prostate. A PSA test measures these levels in a man's blood.
  ng/ml | 2.3 (2.4) | 0.6 (0.8) | 2.0 (2.3)
Qmax (Free Flow Study) [Mean (Standard Deviation); unit: ml/sec] — Maximum flow rate (Qmax) is the the maximum recorded flow rate
  ml/sec | 9.3 (5.2) | 12.4 (6.6) | 10.0 (5.5)
Voided Volume (Free Flow Study) [Mean (Standard Deviation); unit: ml] | 173 (92) | 299 (230) | 197 (134)
Postvoid residual volume (PVR) (Free Flow Study) [Mean (Standard Deviation); unit: ml] — Postvoid residual volume (PVR) is the volume of fluid remaining in the bladder immediately after the completion of micturition.
  ml | 162 (206) | 157 (113) | 161 (188)
Qmax (Pressure flow study) [Mean (Standard Deviation); unit: ml/sec] | 5.7 (3.7) | 10.4 (5.0) | 6.7 (4.4)
Voided Volume (Pressure flow study) [Mean (Standard Deviation); unit: ml] | 150 (104) | 283 (171) | 179 (131)
Postvoid Residual Volume (PVR) (Pressure flow study) [Mean (Standard Deviation); unit: ml] — Measure Description: Postvoid residual volume (PVR) is the volume of fluid remaining in the bladder immediately after the completion of micturition.
  ml | 292 (213) | 270 (209) | 287 (209)
Pdet at Qmax (Pressure flow study) [Mean (Standard Deviation); unit: cm H2O] — Pdet is detrusor pressure at maximum flow rate (Qmax)
  cm H2O | 83 (24) | 33 (13) | 72 (31)
Max Detrusor pressure (Pdet) (Pressure flow study) [Mean (Standard Deviation); unit: cm H2O] — Detrusor pressure (Pdet) -- is that component of vesical pressure that is created by forces in the bladder wall (passive and active).
  cm H2O | 90 (29) | 43 (12) | 80 (32)
Bladder Outlet Obstruction (BOO) Index (Pressure flow study) [Mean (Standard Deviation); unit: units on a scale] — BOOI is a mathematical index of out-let resistance used to help in the diagnosis of men with Benign Prostatic Hyperplasia. Higher values represent an increased amount of bladder outlet obstruction.
  units on a scale | 78 (28) | 16 (10) | 64 (36)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Downward/Flat/Upward Patterns as Assessed by Near Infrared Spectroscopy (NIRS) for BOO Diagnosis
Description: The correlation of the NIRS pattern itself (independent of Qmax and PVR) to BOO. We looked at if the use of the NIRS is a comparable predictor for BOO in patients who were obstructed and those who weren't. The goal of the NIRS is to provide a non-invasive means to diagnose BOO. According to the NIRS algorithm, a downward NIRS pattern related to a higher probability of obstruction and and upward pattern relates to a higher probability of non obstruction.
Time Frame: Assessed at 3 and 6 months, post operatively
Measure: Number; unit: participants
Groups:
- Number Obstructed; Number Unobstructed: Free Flow and pressure flow NIRS patterns
- Totals: Total number of participants included
Arm/Group | Number Obstructed | Number Unobstructed | Totals
Number analyzed (Participants) | 26 | 7 | 33
participants
  Free Flow NIRS Downward | 9 | 4 | 13
  Free Flow NIRS Flat | 4 | 1 | 5
  Free Flow NIRS Upward | 13 | 2 | 15
  Pressure Flow NIRS Downward | 11 | 3 | 14
  Pressure Flow NIRS Flat | 2 | 0 | 2
  Pressure Flow NIRS Upward | 5 | 2 | 7

ADVERSE EVENTS:
Groups:
- Obstructed: Those with BOO
- Unobstructed: Those without BOO
Arm/Group | Obstructed | Unobstructed
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/7
Other Adverse Events (participants affected / at risk) | 0/26 | 0/7

LIMITATIONS AND CAVEATS:
Study limitations include sample size and the lack of a control group without LUTS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No